CLINICAL TRIAL: NCT07173933
Title: A Multicenter, Open-label, Single-dose, Dose-escalation Phase I/II Clinical Trial Evaluating the Safety, Tolerability, and Efficacy of GC310 Adeno-associated Virus Injection in the Treatment of Patients With Wilson's Disease (WD)
Brief Title: Phase I/II Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of GC310 Injection in Patients With Wilson's Disease (WD)
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GeneCradle Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JLJY-GC310-WD-001
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Wilson Disease
Keywords: gene therapy; Genecradle; AAV5; ATP7B; Wilson Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Single intravenous administration of GC310 at a dose of 3.0E+13 d.vg/kg
  Interventions: Genetic: GC310
- Cohort 2 (Experimental): Single intravenous administration of GC301 at a dose of 6.0E+13 d.vg/kg
  Interventions: Genetic: GC310

INTERVENTIONS:
Genetic: GC310 — GC310 is an adeno-associated virus 5 (AAV5) vector delivering a functional copy of the truncated human ATP7B gene

SUMMARY:
The goal of this clinical trial is to learn if GC310 (AAV5-ATP7B) gene therapy can treat Wilson's Disease (WD) in patients over the age of 18 years old. The main questions it aims to answer are:

Is GC310 safe and tolerable to WD patients? What is the recommended phase II dose (RP2D)? What is the change from baseline in 24-hour urinary copper concentration after 52 weeks of administration?

Participants will be administrated GC310 intravenously and be followed up for 52 weeks to observe drug safety, tolerability and efficacy .

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years, sex unrestricted;
* Definitive diagnosis of Wilson disease (WD) based on:

  (i) or (ii) + (iii) and (iv), or (i) or (ii) + (v); (i) Neurological and/or psychiatric symptoms; (ii) Unexplained liver injury; (iii) Reduced serum ceruloplasmin and/or elevated 24-hour urinary copper; (iv) Positive corneal Kayser-Fleischer (K-F) ring; (v) Biallelic pathogenic ATP7B variants confirmed by segregation analysis and variant pathogenicity assessment;
* Serum ceruloplasmin concentration < ½ × lower limit of normal (LLN);
* Willing and able to comply with all study procedures, and has provided written informed consent.

Exclusion Criteria:

Subjects meeting ANY of the following criteria will be excluded:

1. Screening serum anti-AAV5 neutralizing antibody titre > 1:100.
2. Clinically significant laboratory abnormality at screening or baseline:

   1. ALT or AST ≥ 5 × ULN, direct bilirubin > 1 × ULN, or albumin < 1 × LLN;
   2. Blood ammonia > 1 × ULN.
3. Renal impairment (any degree).
4. Current hepatic decompensation or history of hepatic decompensation.
5. Liver stiffness measurement (LSM) ≥ 15 kPa by transient elastography at screening.
6. History of acute liver failure from any cause.
7. Evidence of advanced liver disease defined by either:

   1. MELD score ≥ 12, or
   2. Child-Pugh score ≥ 7.
8. Severe neuro-psychiatric manifestations that, in the investigator's opinion, could compromise subject safety or interfere with study participation.
9. Positive for HIV antibody, hepatitis C antibody, Treponema pallidum antibody, or hepatitis B surface antigen.
10. Contraindications to glucocorticoid therapy judged by the investigator (e.g., uncontrolled hypertension, systemic fungal infection, glaucoma, osteoporosis, active tuberculosis).
11. Concurrent conditions that may interfere with study conduct or assessment, including significant gastrointestinal, cardiovascular, cerebrovascular, renal, endocrine, haematological, immunological, neurological or psychiatric disorders other than Wilson disease.
12. Pregnant or lactating women.
13. Women of child-bearing potential or fertile men who plan to conceive within 1 year after dosing or are unwilling to use highly effective contraception.
14. Body-mass index ≥ 24 kg/m².
15. History of severe hypersensitivity to foods or drugs, including recombinant proteins.
16. Vaccination within 2 weeks prior to planned dosing.
17. Prior exposure to any gene-therapy product.
18. Participation in any other clinical trial (WD-related or not) within 3 months before screening.
19. Any other condition or circumstance that, in the opinion of the investigator, renders the subject unsuitable for the study (e.g., poor compliance).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events after GC310 administration | within 12 weeks
Incidence of dose-limiting toxicity (DLT) events after GC310 administration; | within 4 weeks
Change from baseline in serum ceruloplasmin (CP) concentration after GC310 administration; | 52 weeks
Change from baseline in 24-hour urinary copper excretion after GC310 administration. | 52 weeks

SECONDARY OUTCOMES:
Change from baseline in the urinary copper-to-creatinine ratio | 52 weeks
Change from baseline in ALT and AST levels | 52 weeks
Change from baseline in hepatic imaging findings | 52 weeks
Change from baseline in Kayser-Fleischer (K-F) rings observed by slit-lamp examination | 52 weeks
Evaluation of adverse-event incidence | 52 weeks
Serum anti-AAV5 and anti-ATP7B antibody levels | 52 weeks
Change in blood GC310 vector genome copy number | 52 weeks
AAV shedding | 52 weeks

OTHER OUTCOMES:
Change from baseline in serum ceruloplasmin (CP) activity | 52 weeks
Change from baseline in relative exchangeable copper (exchangeable copper/total serum copper) | 52 weeks
Change from baseline in brain MRI findings | 52 weeks
Change from baseline in liver biopsy findings | 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided